CLINICAL TRIAL: NCT05010291
Title: Behavioural Text Messaging to Improve Retention in Care for Patients on Antiretroviral Therapy in Ekurhuleni District, South Africa
Brief Title: Behavioural Text Messages to Improve Retention in Care in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Witwatersrand, South Africa (Other); Aurum Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 210308
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: HIV/AIDS
Keywords: Behavioral sciences; Retention in care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of Care (SOC) messaging (Experimental): Participants randomized into this arm will receive standard voice call reminders + the Standard of Care (SOC) text message reminders. The study team will send these one-way text messages to recipients of care as a reminder 1) approximately 3-7 days in advance of a clinic appointment, or 2) to follow-up approximately 24 hours after a missed clinic appointment. These text messages will include the SOC text
  Interventions: Behavioral: Standard of Care (SOC) text message reminder to attend clinic appointment
- Loss aversion messaging (Experimental): Participants randomized into this arm will receive standard voice call reminders + loss aversion text message reminders. The study team will send these one-way text messages to recipients of care as a reminder 1) approximately 3-7 days in advance of a clinic appointment, or 2) to follow-up approximately 24 hours after a missed clinic appointment. These text messages will include loss aversion framing.
  Interventions: Behavioral: Loss aversion framed text message reminder to attend clinic appointment
- Social norms messaging (Experimental): Participants randomized into this arm will receive standard voice call reminders + social norms text message reminders. The study team will send these one-way text messages to recipients of care as a reminder 1) approximately 3-7 days in advance of a clinic appointment, or 2) to follow-up approximately 24 hours after a missed clinic appointment. These text messages will include social norms framing.
  Interventions: Behavioral: Social norms framed text message reminder to attend clinic appointment
- Altruism messaging (Experimental): Participants randomized into this arm will receive standard voice call reminders + altruism text message reminders. The study team will send these one-way text messages to recipients of care as a reminder 1) approximately 3-7 days in advance of a clinic appointment, or 2) to follow-up approximately 24 hours after a missed clinic appointment. These text messages will include altruism framing.
  Interventions: Behavioral: Altruism framed text message reminder to attend clinic appointment

INTERVENTIONS:
Behavioral: Standard of Care (SOC) text message reminder to attend clinic appointment — SOC one-way text message reminding recipient of care to either 1) attend a scheduled clinic appointment or 2) visit the clinic after a missed appointment.
  Arms: Standard of Care (SOC) messaging
Behavioral: Loss aversion framed text message reminder to attend clinic appointment — Loss aversion framed one-way text message reminding recipient of care to either 1) attend a scheduled clinic appointment or 2) visit the clinic after a missed appointment.
  Arms: Loss aversion messaging
Behavioral: Social norms framed text message reminder to attend clinic appointment — Social norms framed one-way text message reminding recipient of care to either 1) attend a scheduled clinic appointment or 2) visit the clinic after a missed appointment.
  Arms: Social norms messaging
Behavioral: Altruism framed text message reminder to attend clinic appointment — Altruism framed one-way text message reminding recipient of care to either 1) attend a scheduled clinic appointment or 2) visit the clinic after a missed appointment.
  Arms: Altruism messaging

SUMMARY:
The proportion of South Africans aware of their HIV status and on treatment remains lower than optimal. The goal of this study is to rapidly determine whether text messages framed according to behavioural economics principles increase clinic attendance among recipients of care on antiretroviral therapy in South Africa. We hypothesize that messages incorporating behavioural economics principles will increase the likelihood of recipients of care attending clinic appointments and returning within 28 days of a missed appointment.

DETAILED DESCRIPTION:
The objective of this study is to rapidly determine whether text messages framed according to behavioural economics principles increase the likelihood that recipients of care attend their clinic appointment and return to clinic within 28 days of a missed appointment. The study will be nested in a routine HIV program, in approximately 5 selected Aurum Institute clinics based in Ekurhuleni district, Gauteng province, South Africa.

Intervention arms will include voice call attempts and one-way text messages sent by clinic staff to recipients of care in two scenarios: 1) Approximately 3-7 days in advance of a clinic appointment for collecting antiretroviral medication supplies or collection of a specimen for viral load testing and 2) Approximately 24 hours after a missed clinic appointment.

This individually randomised trial will have four arms. Each time there is an upcoming or missed clinic visit clinic staff will randomly assign recipients of care to one of the following study arms: 1) Standard of Care 2) Loss aversion framed messaging 3) Social norms framed messaging or 4) Altruism framed messaging.

ELIGIBILITY:
Inclusion Criteria:

* Registered to receive ART (this includes patients receiving ART through multi-month scripting) at selected study sites.
* Aged ≥18 years.
* Have a documented cell phone number in their clinic records
* Are eligible to receive appointment reminders as part of routine care OR eligible to receive follow-up text messages as part of routine care for missed clinic appointments.

Exclusion Criteria:

* Do not have contact details in their clinic records.
* Have contact details on record that are established to belong to someone else upon follow-up (i.e., wrong number).
* Have contact details that are deactivated/non-functional (i.e., voice notification that the number does not exist).
* Are documented to have self-transferred out of the clinic.
* Are known to have been deceased.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1541 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Appointment reminders | Approximately 3-5 months
  Proportion of clients with schedule clinic visit attendance, defined as the number of patients with a verified clinic on the scheduled appointment day/the total number of clients that were sent appointment reminders (stratified by study arm).
Missed clinic appointments | Approximately 3-5 months
  Proportion of patients with a verified clinic visit within 28 days of missing a scheduled clinic appointment defined as the number of patients with a verified clinic within 28 days of missing a scheduled clinic appointment/the total number of clients that Tracers sent text messages following a missed clinic appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Tonderai Mabuto, PhD, Principal Investigator — Aurum Institute; Harsha Thirumurthy, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Aurum Institute, Johannesburg, Gauteng, South Africa